CLINICAL TRIAL: NCT05172882
Title: Comparison of the Efficacy of Transversalis Fascia Plane Block and Wound Infiltration in Varicoselectomy Surgery; Randomised, Controlled Study.
Brief Title: Efficacy of Transversalis Fascia Plane Block Versus Wound Infiltration in Varicoselectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Erkan Cem ÇELİK, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATATÜRK ÜNİVERSİTESİ
Record Dates: First submitted 2021-11-23; First posted 2021-12-29 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Analgesia; Transversalis Fascia Plane Block; Wound Infiltration; Varicoselectomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wound Infiltration (Experimental): Wound infiltration will be applied to the surgical incision site for patients in this group. Infiltration fluid will contain 20 ml 0.25% bupivakain.
  Interventions: Procedure: Wound site infiltration
- Transversalis Fascia Plane Block (Experimental): Transversalis fascia plane block will be performed on only one periinguinal side for patients in this group. Block fluid will contain 20 ml 0.25% bupivakain.
  Interventions: Procedure: Transversalis fascia plane block

INTERVENTIONS:
Procedure: Wound site infiltration — Block fluids that were prepared as 20 ml 0.25% bupivacaine before the intervention, will be applied through the upper and lower incision lips on the suprainguinal surgical site.
  Arms: Wound Infiltration
Procedure: Transversalis fascia plane block — External, internal oblique, and transversus abdominis muscles will be visualized by the ultrasound device. After transversalis fascia will be seen, transversalis fascia plane block will be performed. As a block fluid 20 ml 0.25% bupivacaine will be applied.
  Arms: Transversalis Fascia Plane Block

SUMMARY:
Before surgery, patients will be divided into 2 groups as transversalis fascia plane block will be applied and skin infiltration will be applied. Post-operative analgesic procedures will be applied to patients receiving general anesthesia. Postoperative analgesic consumption and pain scores of the patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who will undergo Varicocele operation
* ASA I-II

Exclusion Criteria:

* Patients with allergic reaction to anesthesia and analgesia drugs to be used
* Patients who did not want to voluntarily participate in the study
* Severe systemic disease (kidney, liver, pulmonary, endocrine)
* Substance abuse history
* Chronic pain history
* Psychiatric problems and communication difficulties
* History of hematological problem
* Patients with severe hemodynamic instability due to infection, heavy bleeding

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Pain Scores (0 (low)-10 (high)) | 1st hour
  Pain will be assessed by visual analog scale scores
Pain Scores (0 (low)-10 (high)) | 2nd hour
  Pain will be assessed by visual analog scale scores
Pain Scores (0 (low)-10 (high)) | 4th hour
  Pain will be assessed by visual analog scale scores
Pain Scores (0 (low)-10 (high)) | 8th hour
  Pain will be assessed by visual analog scale scores
Pain Scores (0 (low)-10 (high)) | 12th hour
  Pain will be assessed by visual analog scale scores
Pain Scores (0 (low)-10 (high)) | 24th hour
  Pain will be assessed by visual analog scale scores

SECONDARY OUTCOMES:
Rescue analgesic consumption | Any time on postsurgical first 24 hour.
  Analgesic drug consumption will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Erkan Cem ÇELİK, Erzurum, Turkey (Türkiye)